CLINICAL TRIAL: NCT00102843
Title: Effect of Lowering of Fasting Plasma Homocysteine Concentrations Through Supplementation With Betaine or Folic Acid on Vascular Function in Healthy Volunteers
Brief Title: Effect of Betaine and Folic Acid on Vascular Function in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen Centre for Food Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: P02.0505L
Record Dates: First submitted 2005-02-03; First posted 2005-02-04 (Estimated); Last update posted 2005-08-03 (Estimated); Status verified 2005-08

CONDITIONS: Healthy; Cardiovascular Diseases
Keywords: folic acid; betaine; homocysteine; cardiovascular disease prevention; human; Cardiovascular health
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements; Folic Acid; Betaine

INTERVENTIONS:
Procedure: supplementation with folic acid and betaine

SUMMARY:
The purpose of this study is to determine whether lowering of fasting homocysteine concentrations improves vascular function in healthy volunteers, irrespective of the homocysteine-lowering agent.

DETAILED DESCRIPTION:
A high plasma homocysteine is a potential risk factor for cardiovascular disease and death. However, it remains uncertain whether homocysteine per se, low status of folate, or other factors related to methionine metabolism are involved in the pathogenesis of cardiovascular disease. Previous studies have shown that a high concentration of homocysteine in blood is related to an impaired vascular function in the arteries, an indicator of cardiovascular disease risk. Virtually all intervention trials used folic acid as a homocysteine-lowering agent, which may however affect vascular function through mechanisms not related to homocysteine. We investigated whether lowering of fasting homocysteine concentrations via supplementation with betaine or folic acid improves vascular function in healthy volunteers, in order to distinguish between effects of folic acid and of homocysteine-lowering per se.

Comparison: We compare the effects of supplementation with folic acid to the effects of betaine, and to the effects of a placebo on plasma homocysteine concentrations and vascular function in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy.
* Women postmenopausal: two or more years after last menstruation. If the uterus was surgically removed, the women must be 55 years or older.
* Normal blood values for: hematology, total homocysteine, blood lipids, vitamin B6, vitamin B12, folate, liver enzymes, creatinine.
* Absence of protein and glucose in urine sample.
* Body mass index (BMI) between 18 and 30 kg/m2.
* Good ultrasound visibility of the brachial artery, judged by the sonographer.
* Willing not to use supplements containing B-vitamins, antioxidant vitamins (A, beta-carotene, C and E) or n-3 fatty acids/fish oil supplements from screening day (>2 months before start of the study) until end of study.
* Willing not to be blood or plasmapheresis donor from 4 weeks before the screening day, and 4 weeks before the start of the study until the end of study.

Exclusion Criteria:

* Any chronic or acute disease (e.g. diabetes, renal disease, inflammation).
* Current, or history of cardiovascular disease.
* Hypertension.
* Medical history or surgical events known to interfere with the study.
* Fasting plasma total homocysteine > 26 micromol/L.
* Alcohol consumption: more than 21 consumptions /week for women, and more than 28 consumptions/week for men.
* Weight loss or gain > 2 kg in the month prior to screening.
* Any special diet (prescribed, slimming, macrobiotic or total vegetarian). Sole exclusion of meat and fish from an otherwise 'normal' western diet is allowed.
* Lactose intolerance.
* Use of supplements containing B-vitamins more than once weekly in the period from 3 months before the screening day.
* Participation in any other trial up to 3 months before this study.
* Use of medication known to interfere with the study outcome.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-10; Study Completion 2003-06

PRIMARY OUTCOMES:
Concentrations of plasma homocysteine in fasting state
Vascular function, measured as flow mediated vasodilation, in fasting state

SECONDARY OUTCOMES:
Lipid concentrations
B-vitamins
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Petra Verhoef, PhD, Study Chair — Wageningen Centre for Food Sciences
Locations (1):
- Wageningen Centre for Food Sciences, Wageningen, Netherlands